CLINICAL TRIAL: NCT06876337
Title: Frequency of Skin Diseases in Children with Inborn Errors of Immunity
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Norhan Gamal El-Deen Mohamed, Assistant Lecturer, Assiut University
Other Study IDs: skin diseases in children IEM
Record Dates: First submitted 2025-03-08; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
1. To detect the prevalence of skin diseases in patients with IEI in Assiut university Children hospital.
2. To describe the pattern of dermatological manifestation among IEI patients present at Assiut University Children hospital.

DETAILED DESCRIPTION:
The immune system is a complex network of cells and organs which cooperate to protect individuals against infectious microorganisms. B- and T- lymphocytes, phagocytic cells, and soluble factors such as complement are some of the major components of the immune system and have specific critical functions in immune defense. When part of the immune system is missing or does not work correctly, immunodeficiency occurs; it may be either congenital (primary) or acquired (secondary). Primary immunodeficiency diseases (PIDs), also known as inborn errors of the immune system (IEI), are a heterogeneous group of inherited disorders caused by genetic mutations that alter the immune system.

Individual IEI are rare, IEIs as a group are not, and they represent a significant health burden. The updated classification of Inborn Errors of Immunity (IEI), encompassing a total of 555 IEIs, and 17 phenocopies due to mutations in 504 different genes. IEIs are currently categorized into 10 categories, with overlapping phenotypes. These categories are Combined immunodeficiencies, Combined immunodeficiencies with syndromic features, Predominantly antibody deficiencies, Diseases of immune dysregulation, Congenital defects of phagocytes, Defects in intrinsic and innate immunity, Autoinflammatory diseases, Complement deficiencies, Bone Marrow Failure, and Phenocopies of inborn errors of immunity.

IEIs present clinically as increased susceptibility to infections, autoimmunity, autoinflammation, allergy, bone marrow failure, and/or malignancy. IEI is to be suspected if there is recurrent or opportunistic infections, organ specific inflammation, autoimmunity, or continuous systemic immune activation and/or benign or malignant, potentially virally induced lymphoproliferation or tumors are seen together, in various combinations.

The skin is an organ of great importance at the immunological level and is commonly affected in IEI. Although infections are the most common cutaneous finding in IEI patients, noninfectious skin diseases are also quite frequent among those patients. These include allergic, inflammatory autoimmune, and malignant manifestations. Also, pigmentary changes, angioedema, urticaria, vasculitis along with nonspecific findings of eczema, erythroderma, granuloma, and ectodermal dysplasia are among the early presenting symptoms in IEI.

Severe combined immunodeficiency (SCID) patients present with severe, recurrent viral and bacterial infections as well as opportunistic infections very early in life (before 6 months of age). IEI is associated with atopy commonly include severe atopic dermatitis as a distinctive characteristic of the disease due to an immune dysregulation that affects skin barrier function.

To the best of our knowledge, data about the cutaneous manifestations of IEI among patients attending Assiut university Children Hospital are lacking. Thus, the goal of this study is to describe the clinical characteristics of the skin manifestations of pediatric patients diagnosed with IEI, this may deepen the knowledge and increase awareness of physicians about alarming cutaneous finding for IEI, aiding in earlier diagnosis and better management of those patient.

ELIGIBILITY:
Inclusion Criteria:

* • Age of patients below 18 years old.

  * Both sexes.
  * Patients diagnosed with IEI according to the clinical and laboratory criteria outlined by the latest International Union of Immunological Societies (IUIS) classification or equivalent recognized diagnostic guidelines.

Exclusion Criteria:

* Patients older than 18 years Patients not fulfilling the criteria for diagnosis of IEI or still not diagnosed yet.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Age of patients below 18 years old. both sex,at the Allergy, Immunology, and Rheumatology Unit of Assiut University Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
detect the prevalence of skin diseases in patients with IEI in Assiut university Children hospital | from march 2025 to february 2026
  To describe the pattern of dermatological manifestation among IEI patients present at Assiut University Children hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Norhan Gamal, Asyut, Egypt

REFERENCES:
- [Background] Al-Herz W, Zainal M, Nanda A. A Prospective Survey of Skin Manifestations in Children With Inborn Errors of Immunity From a National Registry Over 17 Years. Front Immunol. 2021 Sep 30;12:751469. doi: 10.3389/fimmu.2021.751469. eCollection 2021. PMID 34659256
- [Background] Kang JM, Kim SK, Kim D, Choi SR, Lim YJ, Kim SK, Park BK, Park WS, Kang ES, Ko YH, Choe YH, Lee JW, Kim YJ. Successful Sirolimus Treatment for Korean Patients with Activated Phosphoinositide 3-kinase delta Syndrome 1: the First Case Series in Korea. Yonsei Med J. 2020 Jun;61(6):542-546. doi: 10.3349/ymj.2020.61.6.542. PMID 32469178
- [Background] Fischer A, Notarangelo LD, Neven B, Cavazzana M, Puck JM. Severe combined immunodeficiencies and related disorders. Nat Rev Dis Primers. 2015 Oct 29;1:15061. doi: 10.1038/nrdp.2015.61. PMID 27189259
- [Background] Cagdas D, Ayasun R, Gulseren D, Sanal O, Tezcan I. Cutaneous Findings in Inborn Errors of Immunity: An Immunologist's Perspective. J Allergy Clin Immunol Pract. 2023 Oct;11(10):3030-3039. doi: 10.1016/j.jaip.2023.06.037. Epub 2023 Jun 28. PMID 37391021
- [Background] Lehman H. Skin manifestations of primary immune deficiency. Clin Rev Allergy Immunol. 2014 Apr;46(2):112-9. doi: 10.1007/s12016-013-8377-8. PMID 23760761
- [Background] Allenspach E, Torgerson TR. Autoimmunity and Primary Immunodeficiency Disorders. J Clin Immunol. 2016 May;36 Suppl 1:57-67. doi: 10.1007/s10875-016-0294-1. Epub 2016 May 23. PMID 27210535
- [Background] de Wit J, Brada RJK, van Veldhuizen J, Dalm VASH, Pasmans SGMA. Skin disorders are prominent features in primary immunodeficiency diseases: A systematic overview of current data. Allergy. 2019 Mar;74(3):464-482. doi: 10.1111/all.13681. Epub 2018 Dec 27. PMID 30480813
- [Background] Subbarayan A, Colarusso G, Hughes SM, Gennery AR, Slatter M, Cant AJ, Arkwright PD. Clinical features that identify children with primary immunodeficiency diseases. Pediatrics. 2011 May;127(5):810-6. doi: 10.1542/peds.2010-3680. Epub 2011 Apr 11. PMID 21482601
- [Background] Arkwright PD, Gennery AR. Ten warning signs of primary immunodeficiency: a new paradigm is needed for the 21st century. Ann N Y Acad Sci. 2011 Nov;1238:7-14. doi: 10.1111/j.1749-6632.2011.06206.x. PMID 22129048
- [Background] Kobrynski L, Powell RW, Bowen S. Prevalence and morbidity of primary immunodeficiency diseases, United States 2001-2007. J Clin Immunol. 2014 Nov;34(8):954-61. doi: 10.1007/s10875-014-0102-8. Epub 2014 Sep 26. PMID 25257253
- [Background] Riaz IB, Faridi W, Patnaik MM, Abraham RS. A Systematic Review on Predisposition to Lymphoid (B and T cell) Neoplasias in Patients With Primary Immunodeficiencies and Immune Dysregulatory Disorders (Inborn Errors of Immunity). Front Immunol. 2019 Apr 16;10:777. doi: 10.3389/fimmu.2019.00777. eCollection 2019. PMID 31057537